CLINICAL TRIAL: NCT03338699
Title: Evaluation of the ShangRing vs. Mogen Clamp for Early Infant Male Circumcision (EIMC) in Sub-Saharan Africa
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Population Council (Other); Johns Hopkins University (Other); Jhpiego (Other); George Washington University (Other); Bill and Melinda Gates Foundation (Other); Rakai Health Sciences Program (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1611017762
Record Dates: First submitted 2017-10-04; First posted 2017-11-09 (Actual); Last update posted 2021-03-04 (Actual); Status verified 2021-02

CONDITIONS: Circumcision
Keywords: Early infant male circumcision; ShangRing; sub-Saharan Africa; HIV; WHO

STUDY DESIGN:
Intervention Model Description: In the pilot phase of the study, participating infants will be allocated to circumcision with either the ShangRing or Mogen clamp. Infants will be randomized in a 1:1 fashion. (Total enrollment: 1380)
  In the second phase of the study, participating infants will receive circumcision with the ShangRing as part of our Field Study design. (Total enrollment: 1690)
  (Total trial enrollment: 3070)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- ShangRing (Experimental): Topical anesthesia based, no-flip ShangRing circumcision.
  Interventions: Device: ShangRing
- Mogen clamp (Active Comparator): Mogen clamp circumcision.
  Interventions: Device: Mogen clamp

INTERVENTIONS:
Device: ShangRing — Topical anesthesia based, no-flip ShangRing circumcision.
  Arms: ShangRing
Device: Mogen clamp — Mogen clamp circumcision
  Arms: Mogen clamp

SUMMARY:
The study will evaluate the safety and acceptability of the topical anesthesia-based, no-flip ShangRing technique vs. Mogen clamp for Early Infant Male Circumcision (EIMC) in neonates and infants up to 60 days of life.

The study will consist of 2 phases; a pilot phase and a field study. In the pilot phase, male infants of up to 60 days of life will be enrolled in three sub-Saharan countries, specifically Kenya, Tanzania, and Uganda. Infants will be randomized in 1:1 fashion to undergo EIMC using either the Mogen clamp or no-flip ShangRing technique using topical anesthesia. Upon completion of the pilot trial and assuming satisfactory safety results, a larger non-comparative field study of ShangRing EIMC will be initiated, as performed by non-physician providers in routine practice settings in the three sub-Saharan African countries.

Total study duration will be 3 years. The pilot phase is anticipated to encompass a total of 1 year. Completion of the field study is expected to take 2 years.

Study Endpoints include:

1. To compare the rates of adverse events (AEs) with the ShangRing or Mogen clamp
2. To compare pain control, time to complete wound healing and parent satisfaction with EIMC using the ShangRing or Mogen clamp
3. To compare operative time and provider preference.
4. To assess the rate of spontaneous ring detachment with the ShangRing as a method to decrease the need for follow-up visits after circumcision.
5. To assess the subpreputial microbiome of the infants prior to and after the initiation of circumcision

Three correlative studies will be conducted:

1. Penile microbiome study: In the pilot trial, the subpreputial microbiome of the infants undergoing circumcision will be assessed to better understand the spectrum of bacteria that may exist and play a role in infant circumcision.
2. Demand creation study: During both the pilot phase and the field study, it will be assessed whether device-driven EIMC can be safely and effectively integrated into maternal and child health services as a method to promote demand creation.
3. Cost impact study: During both the pilot phase and the field study, a comparative cost analysis of EIMC with ShangRing versus Mogen clamp will be performed, in addition to a cost analysis of ShangRing EIMC as performed in routine clinical settings in the field study. The costing of demand creation will also be assessed.

DETAILED DESCRIPTION:
Male circumcision (MC) has been shown to reduce HIV incidence in men by 50-60% in three randomized trials, and observational studies of men circumcised in infancy or childhood have shown long-term protection from HIV acquisition in adulthood. MC also reduces the risk of human papilloma virus, herpes simplex virus type 2 in men; and Trichomonas vaginalis and bacterial vaginosis infections in their female partners, genital ulcer disease in both sexes, and reduces the risk of cervical and penile cancers. In children, circumcision also provides immediate benefits by protecting against urinary tract infections, phimosis, and balanitis.

Though HIV prevention may be achieved through continued scale-up of MC in adolescents and adults, long-term sustainability will likely be better achieved through early infant male circumcision (EIMC). EIMC is technically simpler, safer, and less expensive compared to MC performed in older children or adults. In addition, EIMC has the benefit of more rapid wound healing and does not carry the risk of premature resumption of sexual activity before complete wound healing that has been reported in 7 to 28% of adult men after circumcision which may increase transmission to female partners. In several African countries, EIMC services have been found to be highly acceptable among parents and other caregivers.The long-term benefits of EIMC have led experts to recommend population-wide neonatal circumcision, as the benefits accrued over a child's life greatly outweigh any short-term risks, and delaying circumcision until adulthood places the child at risk of disease acquisition before the procedure can be performed. Despite these advantages, however, EIMC has not been significantly deployed in African countries. Part of the barrier to wider use of EIMC stems from the scarcity of trained providers and resources in sub-Saharan Africa. Device-assisted MC has therefore been proposed to simplify the procedure, enable safe task-shifting, and reduce the burden on healthcare providers, thus increasing the availability of EIMC services. While several devices are currently in use for patients of various ages, the use of a single device requiring only topical anesthesia across all age ranges would dramatically simplify supply chain logistics, streamline personnel training, and most importantly enhance patient/parent acceptability and demand uptake.

This study seeks to accomplish three major goals. First, the study would evaluate the safety of the ShangRing vs. the Mogen clamp for EIMC. The ShangRing is the only MC device requiring topical anesthesia that is capable of being used across all age ranges from newborns to adults; its use would dramatically simplify supply chain logistics, streamline personnel training, and most importantly enhance patient/parent acceptability and demand uptake. The Mogen clamp is a pre-existing device already in use for EIMC in Africa and will serve as an important comparator. The use of an EIMC device that enables safe task-shifting would allow the integration of circumcision services into pre-existing maternal and child health (MCH) service infrastructure and would thereby further facilitate rapid scale-up of MC services throughout Africa. A penile microbiome study will also be performed to better understand the spectrum of bacteria present at the time of EIMC. Next, the study attempts to ascertain whether device-driven EIMC can be safely and effectively integrated into MCH services as a method to promote demand creation. As sub-Saharan countries have deployed MC services on a national basis, the issue of insufficient patient demand has begun to take greater prominence as a barrier to achieving the goal of 20.8 million MC as proposed by the World Health Organization (WHO) and the Joint United Nations Program on HIV/AIDS (UNAIDS). The study will therefore examine the ability of EIMC to stimulate demand for circumcision through MCH services as well as identify potential barriers and strategies for wider scale programmatic roll-out. Finally, the study will also attempt to assess the economic burden of device-driven EIMC. In a context of limited resources, understanding the economic burden of a device-driven EIMC program will be critical in ascertaining its long-term feasibility and sustainability in sub-Saharan Africa.

All subjects will be recruited for the study at the following designated study sites:

Kenya: Homa Bay County Teaching and Referral Hospital, Homa bay; Jaramaogi Oginga Odinga Teaching and Referral hospital, Kisumu County; Nyanza Reproductive Health Society - UNIM Research and Training Centre (URTC) on the grounds of the Lumumba sub-County Hospital, Kisumu County.

Tanzania: Iringa Regional Referral Hospital, Iringa; Ilulu Hospital, Ilula; Mafinga Hospital, Mafinga; Ngome Health Center, Iringa.

Uganda: Rakai District Hospital, Rakai; Kalisizo Hospital, Kyotera; Kakuuto Health Centre IV, Kyotera; Lyantonde District Hospital, Lyantonde, Masaka Regional Referral Hospital, Masaka.

Subjects will be registered to take part in the study through their parents/legally acceptable representatives (LARs) who will be required to sign an informed consent after they agree to the enrollment of their infant. Parents/LARs are first familiarized with the procedures and provided with the information on the risks and benefits of EIMC using WHO/JHPIEGO guidelines.

Each infant will be enrolled in this study for a total of 42 days in the pilot phase and 28 days in the field study (or longer if wound healing is incomplete). Circumcision will take place on day 0, and weekly follow-up visits will be conducted until complete wound healing is documented for the pilot study. For the field study, follow-up will occur on days 7 and 28 only, with additional follow up visits if complete wound healing has not been achieved.

Participation in this study is voluntary. Any parent/LAR is free to discontinue their infant's participation at any point in time. When further participation in the study is not desired, even while the ring is still on, treatment will be administered as if the infant was in the study. However, participation for the entire length of the study is encouraged until the infant is fully healed.

The study doctor or his designee can stop an infant's participation in a study if:

* Continuing in the study could harm the infant
* The study is stopped.

Clinical data will be obtained and recorded using either 1) electronic Clinical Research Forms (eCRFs) that are loaded on mobile tablets or 2) paper forms. The information that will be obtained includes questionnaires, medical history, physical exam findings, details of the EIMC procedure, and clinical follow-up parameters. Once an eCRF is completed, the data will be encrypted on the collecting devices and submitted through a secure connection to the database server. No copy of the information will be left on the electronic device after it has been transferred to the database server. This will ensure that there will be no risk of unauthorized access to the data even in the case of device misplacement. All devices that will be used to collect data shall, upon completion of the day's activity, be locked in the study cabinets in a locked room. All electronic data will be backed-up on paper, and security will be ensured by storing the data in a locked cabinet. Data access will only be provided to primary researchers or their designees, and the data set will only be used for the research question asked.

Informed consent forms and participant contact information will not be obtained using electronic media but will instead be obtained using written forms that will be stored in locked cabinets at the study sites.

-Pilot Phase A total sample size of 460 eligible infants in Kenya, 460 eligible infants in Uganda, and 460 eligible infants in Tanzania will be enrolled, assuming successful recruitment and follow-up of a total of 1200 (87%) patients, or 400 patients per country. The anticipated accrual rate is 115 infants per month across the three countries. Infants will be randomized in a 1:1 fashion using a randomization software to EIMC with the ShangRing or the Mogen clamp, resulting in 200 infants receiving ShangRing circumcision and 200 receiving Mogen clamp per site.

This sample size exceeds the recommendations from the World Health Organization for the comparative trial component of the clinical evaluation of MC devices, which is based on an ability to rule out an adverse event (AE) rate of about 5% or more with a new use of a device that has already been shown to be previously safe in a larger group of men in randomized controlled trials (RCTs) and demonstration studies. The primary endpoint will be safety as determined by the rate of moderate to severe AEs using an intention to treat analysis.

Sample size justification: The goal of this study is to determine if the AE rate using ShangRing is not inferior to that for Mogen clamp. The control arm is the Mogen clamp and the anticipated moderate/severe AE rate is 2%. It is felt that the benefits of ShangRing in terms of convenience and acceptability will allow a non-inferiority margin of 2% (absolute). A sample size of 1200 infants (600 per arm), with one formal interim analysis for futility, has approximately 80% power with a (one-sided) alpha = 0.05. The null hypothesis for the non-inferiority test is that the moderate/severe AE rate for the ShangRing is at least 2% (absolute) greater than that of Mogen clamp, which is assumed to be 2%. The alternative hypothesis is that the rate of the ShangRing is less than 2% great than that of the Mogen clamp.

-Field Study The WHO recommends that the field study component of clinical assessment involve at least 500 clients per country in two countries of intended use. As such, we will aim to recruit a maximum of 600 infants in Kenya, 600 infants in Uganda and 600 infants in Tanzania, assuming successful recruitment and follow-up of a total of 1500 (83%) patients, or 500 patients per country. Once a total of 500 infants have completed follow up in each country, recruitment will stop as the necessary sample size will then had been achieved.

Sample size justification: A sample size of 1500 patients will have a 95% confidence interval margin-of-error of 0.007 to 0.010 for the moderate/severe AE rate estimate, assuming the observed rate is between 0.02 and 0.04. This provides adequate precision for the estimate of the severe AE rate in order to make decisions as to whether this device is safe when used in the field.

AEs will be pre-specified based on WHO/JHPIEGO definitions of the nature and severity of AEs, and classified as related or unrelated to EIMC.

-Statistical considerations and data analysis AE rates, pain control, wound healing, and parent/provider satisfaction between groups will be compared using chi-square tests, two-group t-tests. If the variable distributions violate the underlying assumptions of these tests, the corresponding non-parametric tests will be used (e.g. Wilcoxon rank sum test, Fisher's exact test). Analyses will be for all sites, and site-specific. Multivariable models will be used to adjust for imbalances in baseline characteristics significant at p<0.10 using logistic regression to estimate adjusted odds ratios of moderate/severe AEs by arm. For outcomes with an incidence <10%, the modified Poisson regression will be used to estimate adjusted prevalence rate ratios.

A formal interim analysis will be conducted after 200 circumcisions have been completed. The analysis will be for futility only. If after 200 infants have been enrolled and followed for 42 days it is found that the (non-inferiority) p-value is 0.97 or greater (corresponding to a z-statistic of 1.91 or greater) the trial will be recommended to stop due to futility.

ELIGIBILITY:
Inclusion Criteria:

1. Male infants from 24 hours up to 60 days of life
2. Gestational age ≥37 weeks
3. Normal birth weight (≥2.5 Kg)
4. No illness requiring medical treatment
5. No penile abnormality requiring surgical repair (e.g. hypospadias, chordee)
6. No family history of bleeding disorders
7. Consent provided by at least one parent/legally acceptable representative (LAR) of the infant

   1. Parent or LAR must be able to understand study procedures and requirements of study participation;
   2. Parent or LAR must agree to return the client to the study site for the full schedule of follow-up visits after his circumcision;
   3. Parent or LAR must have a cell phone or access to a cell phone

Exclusion Criteria:

* Not meeting one or more of the inclusion criteria
* Consent not provided by parents/legally acceptable representatives of the infant
* If parent(s)/legally acceptable representative(s) decline(s) the procedure or is/are uncomfortable with the procedure
* Babies <6 weeks of age to mother without previous T.T. vaccination during ANC visits for that pregnancy
* Babies >6 weeks of age without DPT vaccination
* Any other valid health-related issues as judged by the health workers

Ages: 24 Hours to 60 Days | Sex: Male | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — All participants in this study are male who will undergo early infant circumcision.
Enrollment: 1380 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Number and severity of adverse events in participants undergoing circumcision with either device based on WHO/JHPIEGO definitions and guidelines. | Up to 8 weeks post-circumcision.
  Adverse events will be pre-specified based on WHO/JHPIEGO definitions of the nature and severity of adverse events, and classified as related or unrelated to EIMC. Adverse events will also include device-related malfunctions and displacements.

SECONDARY OUTCOMES:
Pain scores associated with the circumcision procedure by either device, assessed using the Neonatal Infant Pain Scale (NIPS). | At the time of circumcision procedure.
  Pain scores will be recorded at the time of circumcision procedure using NIPS. NIPS is based on facial expression, crying, breathing patterns, movement of arms and legs, and state of arousal of the infant. A score of 0 is classified as no pain while a score of 6 is most severe.
Time to complete wound healing based on having an intact clean scar with no dehiscence. | Till complete wound healing is reported, up to 8 weeks post-circumcision.
  Circumcision wound is examined at each follow-up visit to check for complete healing. Additional follow-up visits may be needed if complete healing was not reported at the end of scheduled visits.
Parent satisfaction based on post-circumcision interviews. | Up to 8 weeks post-circumcision.
  Parents will be interviewed after their infant had undergone circumcision to express their views on the procedure. They will be required to note whether they are satisfied or dissatisfied about different aspects relating to the procedure and the study.
Operative time measured in minutes. | At the time of circumcision on procedure day.
  Providers will record, in minutes, the amount of time required to complete the circumcision procedure with the ShangRing and Mogen clamp. Recorded time will not include duration of anesthesia administration, or duration for the anesthetic to take effect.
Provider preference of circumcision device based on post-circumcision interviews. | Up to 8 weeks post-circumcision.
  Health providers who will perform the circumcision procedures using the ShangRing and Mogen clamp will be interviewed to express their views and degree of satisfaction with the devices.
Spontaneous detachment as a measure to decrease the need of follow-up visits based on the amount of time, in days, it takes for the device to fall off on its own. | Up to 4 weeks post-circumcision.
  Parents/LARs of infants who underwent ShangRing circumcision will be asked about the date of device detachment if the device is no longer attached at the time of visit.

CONTACTS AND LOCATIONS:
Overall Officials: Richard K Lee, MD, MBA, Principal Investigator — Weill Medical College of Cornell University; Philip S Li, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (3):
- Homa Bay County Teaching and Referral Hospital, Homa Bay, Kenya
- Iringa Regional Referral Hospital, Iringa, Tanzania
- Rakai Health Sciences Program, Kalisizo, Rakai, Uganda

IPD SHARING:
Plan to Share IPD: No
Individual participant data will only be shared among study investigators and authorized personnel at the designated study sites. IPD will not be shared with anyone not involved in the design, planning, or execution of the study.

REFERENCES:
- [Background] Bailey RC, Moses S, Parker CB, Agot K, Maclean I, Krieger JN, Williams CF, Campbell RT, Ndinya-Achola JO. Male circumcision for HIV prevention in young men in Kisumu, Kenya: a randomised controlled trial. Lancet. 2007 Feb 24;369(9562):643-56. doi: 10.1016/S0140-6736(07)60312-2. PMID 17321310
- [Background] Gray RH, Kigozi G, Serwadda D, Makumbi F, Watya S, Nalugoda F, Kiwanuka N, Moulton LH, Chaudhary MA, Chen MZ, Sewankambo NK, Wabwire-Mangen F, Bacon MC, Williams CF, Opendi P, Reynolds SJ, Laeyendecker O, Quinn TC, Wawer MJ. Male circumcision for HIV prevention in men in Rakai, Uganda: a randomised trial. Lancet. 2007 Feb 24;369(9562):657-66. doi: 10.1016/S0140-6736(07)60313-4. PMID 17321311
- [Background] Auvert B, Taljaard D, Lagarde E, Sobngwi-Tambekou J, Sitta R, Puren A. Randomized, controlled intervention trial of male circumcision for reduction of HIV infection risk: the ANRS 1265 Trial. PLoS Med. 2005 Nov;2(11):e298. doi: 10.1371/journal.pmed.0020298. Epub 2005 Oct 25. PMID 16231970
- [Background] Tobian AA, Kigozi G, Wawer MJ, Serwadda D, Quinn TC, Gray RH. Herpes simplex virus type-2 assay specificity and male circumcision to reduce herpes simplex virus type-2 acquisition. AIDS. 2013 Jan 2;27(1):147-9. doi: 10.1097/QAD.0b013e32835aa181. PMID 23221430
- [Background] Tobian AA, Serwadda D, Quinn TC, Kigozi G, Gravitt PE, Laeyendecker O, Charvat B, Ssempijja V, Riedesel M, Oliver AE, Nowak RG, Moulton LH, Chen MZ, Reynolds SJ, Wawer MJ, Gray RH. Male circumcision for the prevention of HSV-2 and HPV infections and syphilis. N Engl J Med. 2009 Mar 26;360(13):1298-309. doi: 10.1056/NEJMoa0802556. PMID 19321868
- [Background] Tobian AA, Gray RH. The medical benefits of male circumcision. JAMA. 2011 Oct 5;306(13):1479-80. doi: 10.1001/jama.2011.1431. No abstract available. PMID 21972310
- [Background] Pintye J, Baeten JM, Manhart LE, Celum C, Ronald A, Mugo N, Mujugira A, Cohen C, Were E, Bukusi E, Kiarie J, Heffron R; Partners PrEP Study Team. Association between male circumcision and incidence of syphilis in men and women: a prospective study in HIV-1 serodiscordant heterosexual African couples. Lancet Glob Health. 2014 Nov;2(11):e664-71. doi: 10.1016/S2214-109X(14)70315-8. Epub 2014 Oct 22. PMID 25442691
- [Background] Tobian AA, Gray RH, Quinn TC. Male circumcision for the prevention of acquisition and transmission of sexually transmitted infections: the case for neonatal circumcision. Arch Pediatr Adolesc Med. 2010 Jan;164(1):78-84. doi: 10.1001/archpediatrics.2009.232. PMID 20048246
- [Background] UNAIDS/WHO/SACEMA Expert Group on Modelling the Impact and Cost of Male Circumcision for HIV Prevention. Male circumcision for HIV prevention in high HIV prevalence settings: what can mathematical modelling contribute to informed decision making? PLoS Med. 2009 Sep;6(9):e1000109. doi: 10.1371/journal.pmed.1000109. Epub 2009 Sep 8. PMID 19901974
- [Background] Binagwaho A, Pegurri E, Muita J, Bertozzi S. Male circumcision at different ages in Rwanda: a cost-effectiveness study. PLoS Med. 2010 Jan 19;7(1):e1000211. doi: 10.1371/journal.pmed.1000211. PMID 20098721
- [Background] Kalichman SC. Neonatal circumcision for HIV prevention: Cost, culture, and behavioral considerations. PLoS Med. 2010 Jan 19;7(1):e1000219. doi: 10.1371/journal.pmed.1000219. PMID 20098515
- [Background] Kigozi G, Gray RH, Wawer MJ, Serwadda D, Makumbi F, Watya S, Nalugoda F, Kiwanuka N, Moulton LH, Chen MZ, Sewankambo NK, Wabwire-Mangen F, Bacon MC, Ridzon R, Opendi P, Sempijja V, Settuba A, Buwembo D, Kiggundu V, Anyokorit M, Nkale J, Kighoma N, Charvat B. The safety of adult male circumcision in HIV-infected and uninfected men in Rakai, Uganda. PLoS Med. 2008 Jun 3;5(6):e116. doi: 10.1371/journal.pmed.0050116. PMID 18532873
- [Background] Hewett PC, Hallett TB, Mensch BS, Dzekedzeke K, Zimba-Tembo S, Garnett GP, Todd PE. Sex with stitches: assessing the resumption of sexual activity during the postcircumcision wound-healing period. AIDS. 2012 Mar 27;26(6):749-56. doi: 10.1097/QAD.0b013e32835097ff. PMID 22269970
- [Background] Mugwanya KK, Whalen C, Celum C, Nakku-Joloba E, Katabira E, Baeten JM. Circumcision of male children for reduction of future risk for HIV: acceptability among HIV serodiscordant couples in Kampala, Uganda. PLoS One. 2011;6(7):e22254. doi: 10.1371/journal.pone.0022254. Epub 2011 Jul 20. PMID 21799805
- [Background] Westercamp N, Bailey RC. Acceptability of male circumcision for prevention of HIV/AIDS in sub-Saharan Africa: a review. AIDS Behav. 2007 May;11(3):341-55. doi: 10.1007/s10461-006-9169-4. Epub 2006 Oct 20. PMID 17053855
- [Background] Plank RM, Makhema J, Kebaabetswe P, Hussein F, Lesetedi C, Halperin D, Bassil B, Shapiro R, Lockman S. Acceptability of infant male circumcision as part of HIV prevention and male reproductive health efforts in Gaborone, Botswana, and surrounding areas. AIDS Behav. 2010 Oct;14(5):1198-202. doi: 10.1007/s10461-009-9632-0. PMID 19924526
- [Background] Waters E, Li M, Mugisa B, Bowa K, Linyama D, Stringer E, Stringer J. Acceptability and uptake of neonatal male circumcision in Lusaka, Zambia. AIDS Behav. 2013 Jul;17(6):2114-22. doi: 10.1007/s10461-012-0297-8. PMID 22968397
- [Background] Young MR, Odoyo-June E, Nordstrom SK, Irwin TE, Ongong'a DO, Ochomo B, Agot K, Bailey RC. Factors associated with uptake of infant male circumcision for HIV prevention in western Kenya. Pediatrics. 2012 Jul;130(1):e175-82. doi: 10.1542/peds.2011-2290. Epub 2012 Jun 18. PMID 22711723
- [Background] Albert LM, Akol A, L'Engle K, Tolley EE, Ramirez CB, Opio A, Tumwesigye NM, Thomsen S, Neema S, Baine SO. Acceptability of male circumcision for prevention of HIV infection among men and women in Uganda. AIDS Care. 2011 Dec;23(12):1578-85. doi: 10.1080/09540121.2011.579939. Epub 2011 Jul 7. PMID 21732902
- [Background] Mavhu W, Hatzold K, Laver SM, Sherman J, Tengende BR, Mangenah C, Langhaug LF, Hart G, Cowan FM. Acceptability of early infant male circumcision as an HIV prevention intervention in Zimbabwe: a qualitative perspective. PLoS One. 2012;7(2):e32475. doi: 10.1371/journal.pone.0032475. Epub 2012 Feb 27. PMID 22384258
- [Background] Jarrett P, Kliner M, Walley J. Early infant male circumcision for human immunodeficiency virus prevention: knowledge and attitudes of women attending a rural hospital in Swaziland, Southern Africa. SAHARA J. 2014;11(1):61-6. doi: 10.1080/17290376.2014.929530. Epub 2014 Jun 24. PMID 24957082
- [Background] Young MR, Bailey RC, Odoyo-June E, Irwin TE, Obiero W, Ongong'a DO, Badia JA, Agot K, Nordstrom SK. Safety of over twelve hundred infant male circumcisions using the Mogen clamp in Kenya. PLoS One. 2012;7(10):e47395. doi: 10.1371/journal.pone.0047395. Epub 2012 Oct 17. PMID 23082162
- [Background] Kankaka EN, Murungi T, Kigozi G, Makumbi F, Nabukalu D, Watya S, Kighoma N, Nampijja R, Kayiwa D, Nalugoda F, Serwadda D, Wawer M, Gray RH. Randomised trial of early infant circumcision performed by clinical officers and registered nurse midwives using the Mogen clamp in Rakai, Uganda. BJU Int. 2017 Jan;119(1):164-170. doi: 10.1111/bju.13589. Epub 2016 Sep 6. PMID 27597563
- [Derived] Posada Calderon L, Basourakos SP, Ballman KV, Ho K, Barone MA, Awori Q, Ouma D, Oketch J, Christensen A, Hellar A, Makokha M, Isangu A, Salim R, Lija J, Gray R, Kiboneka S, Anok A, Kigozi G, Nakabuye R, Ddamulira C, Odiya S, Goldstein M, Li PS, Lee RK. Safety and efficacy of the ShangRing for early infant male circumcision in the routine clinical setting. BMJ Glob Health. 2025 Sep 25;10(9):e017903. doi: 10.1136/bmjgh-2024-017903. PMID 40998526
- [Derived] Basourakos SP, Nang QG, Ballman KV, Al Awamlh OAH, Punjani N, Ho K, Barone MA, Awori QD, Ouma D, Oketch J, Christensen AE, Hellar A, Makokha M, Isangu A, Salim R, Lija J, Gray RH, Kiboneka S, Anok A, Kigozi G, Nakabuye R, Ddamulira C, Mulooki A, Odiya S, Nazziwa R, Goldstein M, Li PS, Lee RK. ShangRing versus Mogen clamp for early infant male circumcision in eastern sub-Saharan Africa: a multicentre, non-inferiority, adaptive, randomised controlled trial. Lancet Glob Health. 2022 Oct;10(10):e1514-e1522. doi: 10.1016/S2214-109X(22)00326-6. PMID 36113534